CLINICAL TRIAL: NCT06423196
Title: Efficacy of Upper Limb Blood Flow Restriction in Handball Players. Randomised Clinical Study
Brief Title: Upper Limb Blood Flow Restriction in Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Floss-Hand
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-05

CONDITIONS: Sports Physical Therapy
Keywords: Handball; Blood flow restriction; Muscle strength; Muscle activation; Upper limbs; Physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Three assessments will be made throughout the study: before the intervention (T0), after the experimental phase (T1) and after a 4-week follow-up period (T2). All variables will be assessed by an evaluator blinded to the assignment of the athletes to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention of the experimental group will consist of performing an exercise protocol after carrying out the blood flow restriction. A total of 6 muscle strength exercises will be performed for the proximal (triceps brachii) and forearm (epitrochlear and epicondylar muscles).
  Interventions: Other: Experimental group
- Control group (No Intervention): Patients included in the control group will continue with their pre-study training and activities, without modifying their routine.

INTERVENTIONS:
Other: Experimental group — In the development of the exercises, the players will mobilise dumbbells of different weights that will be estimated according to the calculation of 30% of 1 RM. This workload with dumbbells is based on previous work where blood flow restriction was used in healthy athletes.
  Arms: Experimental group

SUMMARY:
Introduction. Blood flow restriction therapy involves the use of an occlusion cuff placed over an extremity resulting in a partial reduction of arterial blood flow and total restriction of venous return.

Objectives. To analyse the efficacy of a physiotherapy intervention using blood flow restriction in improving upper limb strength in adult handball players.

Methods. Randomised, single-blind, clinical study. 20 athletes will be recruited and randomly assigned to the experimental and control groups. The intervention of the experimental group will consist of performing an exercise protocol after blood flow restriction. The intervention period will last 4 weeks, with a periodicity of 2 weekly sessions of 30 minutes each. The primary variable will be the strength of the triceps, epicondyle and epitrochlear musculature (pressure hand dynamometer). The secondary variable will be the muscle activation of this musculature (surface electromyography).

ELIGIBILITY:
Inclusion Criteria:

* Athletes over 18 years of age.
* Federated in handball at the time of the study.
* No lower limb injuries in the three months prior to the study.
* Signing the informed consent document.

Exclusion Criteria:

* Athletes who have undergone surgery in the year prior to the study.
* People who do not attend at least 80% of the treatment sessions.
* Players who are receiving physiotherapy treatment in parallel to the physical preparation of the team they are playing for.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Assess the muscle strength at screening visit | Screening visit, within the first seven days after treatment and after four weeks follow-up
  Muscle strength will be assessed with a pressure dynamometer (Lafayette Manual Muscle model). The strength of the triceps brachii, epicondyle and epitrochlear musculature will be measured. The evaluation protocol used by Morin et al. will be used. The unit of measurement is the Newton (the higher the value, the greater the muscle strength). The measurements are taken bilaterally. The mean value of the 2 measurements taken shall be used as a measure.

SECONDARY OUTCOMES:
Assess the muscle activation at screening visit | Screening visit, within the first seven days after treatment and after four weeks follow-up
  Muscle activation will be measured by surface electromyography (model SHIMMMER2, Shimmer, Ireland). Electrode placement will be marked on standing subjects, and will be positioned according to European recommendations for the use of surface electromyography. A bipolar SEMG system will be used with circular electrodes of 10 mm diameter, 20 mm apart, placed longitudinally, in the direction of the muscle fibres under study, and with a reference electrode at a distance. The unit of measurement is µV, where the higher the score, the greater the muscle activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided